CLINICAL TRIAL: NCT04790474
Title: A Single-arm, Multisite, Prospective Study of Ixazomib-pomalidomide-dexamethasone as Second or Third-line Combination Treatment for Patients With Relapsed and Refractory Multiple Myeloma (RRMM) Previously Treated With Daratumumab, Lenalidomide and Bortezomib (IPoD-790 Study)
Brief Title: Ixazomib-pomalidomide-dexamethasone as Second or Third-line Combination Treatment for Patients With Relapsed and Refractory Multiple Myeloma Previously Treated With Daratumumab, Lenalidomide and Bortezomib
Acronym: IPoD-790
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0776-19-TLV
Record Dates: First submitted 2021-03-07; First posted 2021-03-10 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma in Relapse; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ixazomib-pomalidomide-dexamethasone as second or third-line combination treatment (Experimental): Prospective study of ixazomib-pomalidomide-dexamethasone as second or third-line combination treatment for patients with relapsed and refractory multiple myeloma (RRMM) previously treated with daratumumab, lenalidomide and bortezomib
  Interventions: Drug: ixazomib-pomalidomide-dexamethasone

INTERVENTIONS:
Drug: ixazomib-pomalidomide-dexamethasone — Cycles 1-3: during each 21-day cycle:
  * ixazomib 3 mg on Days 1, 4, 8 and 11
  * pomalidomide 4 mg on Days 1 through 14
  * dexamethasone 20 mg on Days 1, 2, 8, 9, 15, 16
  Cycle 4 and consequently: during each 28-day cycle:
  * ixazomib 4 mg on Days 1, 8 and 15
  * pomalidomide 4 mg on Days 1 through 21
  * dexamethasone 20 mg on Days 1, 2, 8, 9, 15, 16, 22 and 23

SUMMARY:
Adult patients with a confirmed diagnosis of symptomatic and relapsed and/or refractory MM, after receiving bortezomib, lenalidomide and daratumumab during first and second lines, will be eligible to be enrolled in this study.

During the first three treatment cycles, patients will be seen twice (Days 1 and 15 of the cycle). Starting from cycle 4 and on, patients will be assessed once per cycle (Day 1), until disease progression, for disease response and progression according to the International Myeloma Working Group (IMWG) criteria. After progression, all patients will be followed for survival; for this purpose, patients will be contacted every 12 weeks until death or termination of the study by the Sponsor.

Patients may continue to receive treatment for 24 months or until disease progression (PD) or unacceptable toxicity, the earlier of the three. Dose modifications may be made based on toxicities. Patients who complete study therapy will continue to receive treatment per standard of care.

DETAILED DESCRIPTION:
This phase 2, open-label, single-arm, prospective, multicenter study will evaluate the safety, tolerability and efficacy of ixazomib-pomalidomide-dexamethasone (IPD) as a second or third-line combination treatment for patients with relapsed and/or refractory multiple myeloma (RRMM) who progressed after receiving bortezomib, lenalidomide and daratumumab during first and second lines. The patient population will consist of adult men and women who have a confirmed diagnosis of MM, who have received two prior lines of therapy, and who meet other outlined eligibility criteria. Following confirmation of eligibility, enrolled patients will be treated with pomalidomide plus dexamethasone as standard of care and will also receive ixazomib as a study drug.

The treatment regimen will involve administration of the following drugs:

Cycles 1-3: during each 21-day cycle:

* ixazomib 3 mg on Days 1, 4, 8 and 11
* pomalidomide 4 mg on Days 1 through 14
* dexamethasone 20 mg on Days 1, 2, 8, 9, 15, 16

Cycle 4 and consequently: during each 28-day cycle:

* ixazomib 4 mg on Days 1, 8 and 15
* pomalidomide 4 mg on Days 1 through 21
* dexamethasone 20 mg on Days 1, 2, 8, 9, 15, 16, 22 and 23 Patients may continue to receive treatment for 24 months or until disease progression (PD) or unacceptable toxicity, the earlier of the three. Dose modifications may be made based on toxicities. Patients who complete study therapy will continue to receive treatment per standard of care.

The main efficacy outcome- Progression Free Survival (PFS) is defined as the time from first dose to the date of the first documented tumor progression or death due to any cause. PFS will be determined by an investigator, based upon laboratory data, as defined by the IMWG criteria.

Secondary Endpoints:Objective response rate (ORR)is defined as the proportion of patients who achieve a best overall response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR), as defined using the IMWG criteria.

Overall Survival (OS) OS is defined as the time between the date of first dose and the date of death due to any cause. OS will be censored on the last date a subject was known to be alive.

Time to Response (TTR) Time to Response is defined as the time from the first dose to the date of the first sCR, CR, VGPR, or PR. TTR will be evaluated for responders Duration of Response (DOR) Duration of Response is defined as the time between the date of first response to the date of the first objectively documented tumor progression as assessed by study steering committee according to modified IMWG criteria or death due to any cause prior to subsequent anti-cancer therapy.

Optional Exploratory Analysis RNA sequencing (by Massive Parallel (MARS)-seq method) of fresh or frozen cluster of differentiation 38+ (CD38+)/CD138+ plasma cells (normal and malignant) in the bone marrow of patients

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria:

1. Male or female patients, 18 years of age or older.
2. Multiple myeloma diagnosed according to standard IMWG criteria
3. Patients must have measurable disease defined by at least one of the following five measurements:

   * Serum M-protein 1 g/dL (10 g/L).
   * Urine M-protein 200 mg/24 hours.
   * Serum free light chain assay: involved free light chain level at least 100 mg/L), provided that the serum free light chain ratio is abnormal.
   * A biopsy proven evaluable plasmacytoma
   * Bone marrow plasmacytosis > 30% of total marrow cells
4. Patients received one or two prior lines of therapy which must have included bortezomib, lenalidomide-and daratumumab.
5. Patients must meet the following clinical laboratory criteria:

   * Absolute neutrophil count (ANC) ≥1,000/mm3 and platelet count≥75,000/mm3. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days of enrollment.
   * Total bilirubin ≤1.5 the upper limit of the normal range (ULN).
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 ULN.
   * Calculated creatinine clearance ≥15 mL/min note: Patients with creatinine clearance of 15-50 mL/min will receive pomalidomide at a reduced dose (3 mg), which may subsequently be increased if well tolerated.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
7. Female patients who:

   * Are postmenopausal for at least 24 months before the screening visit, OR
   * Are surgically sterile, OR
   * Who are of childbearing potential, and agree to practice two effective methods of contraception (1 highly effective method and 1 additional effective method) AT the same time, from the time of signing the informed consent through 90 days after the last dose of study treatment, OR agree to completely abstain from heterosexual intercourse, AND
   * Must also adhere to the guidelines of the pomalidomide pregnancy prevention program Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 milli International Units /mL (milli international units) within 10 to 14 days of initiation of Cycle 1 and again within 24 hours of starting Cycle 1. FCBP must also agree to ongoing pregnancy testing. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
8. Male patients, even if surgically sterilized (i.e., status postvasectomy), who:

   * Agree to completely abstain from heterosexual intercourse, OR
   * Agree to practice effective barrier contraception (i.e., latex condom) during sexual contact with a FCBP, even if they have had a successful vasectomy, throughout the entire study treatment period and through 4 months after the last dose of study treatment AND
   * Must also adhere to the guidelines of the pomalidomide pregnancy prevention program.
9. Must be able to take concurrent aspirin 100mg daily (or enoxaparin 40 mg subcutaneously daily [or its equivalent] if allergic to aspirin) as prophylactic anticoagulation.
10. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
11. Patient is willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion criteria:

Patients meeting any of the following exclusion criteria are not eligible to participate in the study:

1. Patient underwent an allogeneic transplantation
2. Female patients who are lactating or pregnant.
3. Major surgery within 14 days before enrollment.
4. Central nervous system involvement
5. Concomitant use of any other antineoplastic treatment with activity against MM (with the exception of ≤40 mg Dexamethasone per day or equivalent for no longer than 4 days).
6. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before enrollment
7. Diagnosis of Waldenstrom's macroglobulinemia, POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes) syndrome, plasma cell leukemia, primary amyloidosis, myelodysplastic syndrome, or myeloproliferative syndrome.
8. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
9. Anti-myeloma therapy as follows prior to screening bone marrow aspiration:

   * Targeted therapy, epigenetic therapy, within 14 days or at least 5 half-lives,whichever is less;
   * Monoclonal antibody treatment for multiple myeloma within 21 days;
   * Cytotoxic therapy within 14 days;
   * Proteasome inhibitor therapy within 14 days;
   * Immunomodulatory agent therapy within 7 days.
   * Radiotherapy within 14 days (with the exception of radiotherapy for spinal cord compression or for pain control that should be discussed and approved by the sponsor- investigator prior to study enrollment). However, if the radiation portal covered ≤5% of the bone marrow reserve, the subject is eligible irrespective of the end date of radiotherapy.
10. Systemic treatment with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of Cytochrome P450, family 3, subfamily A- clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole or strong Cytochrome P450, family 3, subfamily A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort within 14 days before enrollment in the study.
11. Ongoing or active systemic infection, active hepatitis B virus infection, active hepatitis C infection, or known human immunodeficiency virus (HIV) positive.
12. Comorbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
13. Psychiatric illness/social situation that would limit compliance with study requirements.
14. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
15. Inability to swallow oral medication, inability or unwillingness to comply with the drug administration requirements, or known GI disease or planned gastrointestinal (GI) procedure that could interfere with the oral absorption or tolerance of treatment.
16. Diagnosed or treated for another malignancy within 2 years before enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
17. Failure to have fully recovered (ie, Grade 1 toxicity) from the reversible effects of prior chemotherapy.
18. Patient has Grade 3 peripheral neuropathy during the screening period.
19. Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial.
20. Patients that have previously been treated with ixazomib or pomalidomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival-PFS | Up to 2 years from last patient enrollment
  The time from first dose to the date of the first documented tumor progression or death due to any cause

SECONDARY OUTCOMES:
Objective Response Rate-ORR | Up to 2 years from last patient enrollment
  Proportion of patients who achieve a best overall response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR), as defined using the IMWG criteria.
Overall Survival-OS | Up to 2 years from last patient enrollment
  The time between the date of first dose and the date of death due to any cause. OS will be censored on the last date a subject was known to be alive.
Time To Response-TTR | Up to 2 years from last patient enrollment
  The time from the first dose to the date of the first sCR, CR, VGPR, or PR. TTR will be evaluated for responders (BOR is either sCR, CR, VGPR, or PR) only.
Duration of Response-DOR- | Up to 2 years from last patient enrollment
  The time between the date of first response to the date of the first objectively documented tumor progression as assessed by study steering committee according to modified IMWG criteria or death due to any cause prior to subsequent anti-cancer therapy

OTHER OUTCOMES:
Optional Exploratory Analysis- RNA sequencing | Up to 2 years from last patient enrollment
  RNA sequencing-by (Massively Parallel) MARS-seq method of fresh or frozen CD38+(cluster of differentiation 38)/CD138+ plasma cells (normal and malignant) in the bone marrow of patients

CONTACTS AND LOCATIONS:
Overall Officials: Yael Cohen, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center; Noa Lavi, MD, Principal Investigator — Rambam Health Care Campus; Moshe Gat, MD, Principal Investigator — Hadassah Ein-Keerm Medical Center; Iuliana Vaxman, MD, Principal Investigator — Rabin Medical Center; Hila Magen, MD, Principal Investigator — Shiba Tel Hashomer Medical Center; Chezi Ganzel, MD, Principal Investigator — Shearei Zedek Medical Center; Evgeni Chubar, MD, Principal Investigator — Emek Medical Center
Locations (7):
- Israel (7):
  - Emek Medical Center, Afula
  - Rambam Medical Center, Haifa
  - Hadassah Ein-Kerem Medical Center, Jerusalem
  - Shearei Zedek Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Tel Hashomer, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No